CLINICAL TRIAL: NCT04169451
Title: Intrauterine Insemination With Letrozole Versus Intrauterine Insemination in Natural Cycle. A Muticenter Randomized Controlled Trial
Brief Title: IUI With Letrozole Versus in Natural Cycle
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: The 1st Affiliated Hospital of Anhui Medical University (Unknown); The 2nd Affiliated Hospital of Hebei Medical University (Unknown); Tianjin Central Hospitalof Gynecology Obstetrics (Unknown); Yunnan1stpeople's hospital (Unknown)
Responsible Party: Principal Investigator, Jie Qiao, Professor, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IUI with/without stimulation
Record Dates: First submitted 2019-11-17; First posted 2019-11-19 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Intrauterine Insemination; Unexplained Infertility
MeSH Terms: interventions — Letrozole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- letrozole group (Experimental): Women will be given IUI treatment with ovarian stimulation with letrozole 5mg/day starting from day 3 of menstrual cycle for 5 days.
  Interventions: Drug: Letrozole
- natural cycle group (No Intervention): Women will be given IUI treatment without ovarian stimulation.

INTERVENTIONS:
Drug: Letrozole — Women will be randomized to the group with ovarian stimulation with letrozole or the group without stimulation.
  Arms: letrozole group

SUMMARY:
Rationale Intrauterine insemination (IUI) is the treatment of first choice for couples with unexplained and mild male factor infertility in many countries, but it is controversial whether ovarian stimulation improves fertility outcomes. In recent retrospectively collected data, we found that in couples with unexplained and mild male factor infertility undergoing IUI, ovarian stimulation with letrozole increased live birth rate as compared to natural cycle IUI without substantially increasing the multiple pregnancy rate. We therefore intend to perform a randomized clinical trial (RCT) on the subject in five reproductive medical centers in different cities in China.

Objective To test the hypothesis that in couples with unexplained or mild male factor infertility scheduled for an IUI program ovarian stimulation with letrozole increases the live birth rate as compared to natural cycle treatment.

Study design Multicenter randomized controlled trial.

Study population Women diagnosed with unexplained or mild male factor infertility scheduled for treatment with IUI.

Intervention Women will be randomized for ovarian stimulation with letrozole or to natural cycle IUI. In the group allocated to ovarian stimulation, women will receive oral tablets letrozole 5 mg daily from cycle day 3 for 5 days. We will treat the couples for 3 cycles, with a time horizon of 4 months.

Main study parameters/endpoints Primary outcome is live birth resulting from conception within 4 months after randomization. Secondary endpoints are clinical pregnancy, multiple pregnancy, miscarriage rates, pregnancy complications, time to pregnancy leading to live birth.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness The strategies compared are already broadly applied in current practice. No additional risks are expected. There is no benefit for participants, but the results may benefit future infertile couples.

ELIGIBILITY:
Inclusion criteria

In order to be eligible to participate in this study, a participating couple must meet all of the following criteria:

* Being diagnosed with unexplained or mild male infertility
* At least one sided tubal patency, established according to local protocol
* Normal or mild impairment of semen quality defined as total motile sperm count (TMSC) no less than 5million, based on at least one recent semen analysis

Exclusion criteria

A potential participant who meets any of the following criteria will be excluded from study participation:

* Woman with double sided tubal pathology
* Women with irregular cycles, PCOS or other endocrine disorders
* Man with impaired semen quality: total motile sperm count (TMSC) less than 5million

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 982 (Estimated)
Dates: Start 2022-09-29 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
live birth rate | 14 months
  Primary outcome is live birth resulting from conception within 4 months after randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Qiao, Study Director — Peking Unversity Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided